CLINICAL TRIAL: NCT05156190
Title: Cluster-randomized Trial of a Novel Bright Classroom and Artificial Light Renovation in the Prevention of Myopia Among Chinese School-going Children
Brief Title: The Impact of Bright Classroom on Myopia
Acronym: IMPACT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Approval for buiding the classroom has not been obtained.
Sponsor: Queen's University, Belfast (Other)
Collaborators: Queen's University (Other); Clearly (Other); Affiliated Eye Hospital of Nanchang University (Other); The Eye Hospital of Wenzhou Medical University (Other); Zhongshan Ophthalmic Center, Sun Yat-sen University (Other); State Key Laboratory of Subtropical Building Science, South China University of Technology (SCUT) (Unknown); MOH Foundation (Unknown); Velux China (Unknown)
Responsible Party: Principal Investigator, Nathan Congdon, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Bright Classrooms-TP; light renovation (Other: Queen's University, Belfast)
Record Dates: First submitted 2021-09-09; First posted 2021-12-14 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Myopia
Keywords: bright classroom, myopia, RCT, China
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bright classrooms with skylight or renovated artificial light (Experimental): Students will study in bright classrooms with either skylight or renovated artificial light with light level of over 1000 lux on school time for three years and vision will be screened annually.
  Interventions: Other: bright classrooms with light level over 1000 lux
- conventional classrooms (No Intervention): Students will study in conventional classrooms with normal light level for three years and vision will be screened annual.

INTERVENTIONS:
Other: bright classrooms with light level over 1000 lux — Grade 2 primary school students at the intervention groups will study in bright classrooms for three years and incidence of myopia will be compared with those in conventional classrooms
  Arms: bright classrooms with skylight or renovated artificial light

SUMMARY:
This trial aims to test the effectiveness and practicality of study in the Bright Classrooms with skylight and artificial light renovation in reducing incident myopia in Chinese primary school children over three years, as compared to children studying in conventional classrooms.

DETAILED DESCRIPTION:
The investigators now propose a cluster-randomized controlled trial of Bright Classrooms to provide a definitive answer as to their effect on the reduction of myopia incidence with the interventions of students studying in bright classroom from skylight and artificial light renovation. The bright classroom trial will be conducted in Jiangxi Province, South-east China via Nanchang University Affiliated Eye Hospital and the artificial light renovation study will be in Zhejiang Province via Eye Hospital, Wenzhou Medical University. Classroom design and build will be supported by leading firm in this space, Velux. If the principal can be proven that such innovative architectural modifications and classroom light renovation successfully prevent myopia, it will provide an evidence-based justification for a broad variety of low-cost retrofits, new build designs and light renovation appropriate for various Chinese settings. These might include larger windows, skylights, artificial lighting and appropriate seating arrangements. Once in place, such architectural and light interventions could benefit children over many years, without extensive and difficult-to-sustain programs of behaviour change. This proof-of-principle project could address a significant global eye health challenge and have significant and sustainable socio-economic impact for China and built environments elsewhere throughout the world.

Schools selected for the trial are: Yifen County: 2 schools, Lichuan County: 2 schools, Yiyang County: 2 schools, Fuliang County: 1 school and Shanggao County: 1 school.

ELIGIBILITY:
Inclusion Criteria:

* Willingness of parents to give consent
* Membership in randomly-selected classes at the selected schools.

Exclusion Criteria:

* Children without consent from their parents will be excluded.
* Children having myopia (myopic spherical equivalent refractive error of <= -0.5D in one or both eyes) at baseline are excluded from the primary analysis, although they will be included in the secondary analyses, so there will be no need to exclude them from continuing to study with their classmates and use the assigned classroom.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
three-year cumulative incidence of myopia | 3 years
  Three-year cumulative incidence of myopia in the Intervention and Control groups (intermediate incidence at one year will also be measured), defined as spherical equivalent (sphere + ½ cylinder) <= -0.5D in either eye, based on the definition used in the Refractive Error Study in Children.

IPD SHARING:
Plan to Share IPD: No
study subjects will be presented by code, and shared with other researchers